CLINICAL TRIAL: NCT06137378
Title: ELOS - Induction Chemotherapy With Docetaxel and Cisplatin Followed by Radiation Compared to Additional PD-1 Inhibition in CPS ≥1 Advanced Laryngeal/Hypopharyngeal Cancer Suitable for Laryngectomy Selected After Early Response Evaluation
Brief Title: European Larynx Organ Preservation Study (ELOS) [MK-3475-C44]
Acronym: ELOS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Leipzig (Other)
Collaborators: University of Göttingen (Other); University of Jena (Other); University of Cologne (Other); University of Ulm (Other); University of Regensburg (Other); Wuerzburg University Hospital (Other); Technical University of Munich (Other); Ernst von Bergmann Hospital (Other); Universitätsmedizin Mannheim (Other); University of Kiel (Other)
Responsible Party: Principal Investigator, Andreas Dietz, Univ.-Prof. Dr. med. Andreas Dietz, Chairman, Clinic of Otolaryngology, Head and Neck Surgery & Dept. Head Medicine and Oral Health, University of Leipzig
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-502751-61-00; 2022-502751-61-00 (Other: European Medicines Agency (CTIS)); P_00432 (Other: Paul-Ehrlich-Institut)
Record Dates: First submitted 2023-11-13; First posted 2023-11-18 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Squamous Cell Carcinoma of Head and Neck; Hypopharyngeal Squamous Cell Carcinoma; Laryngeal Squamous Cell Carcinoma Stage III; Laryngeal Squamous Cell Carcinoma Stage IV; Squamous Cell Carcinoma of Larynx; Squamous Cell Carcinoma of the Larynx; Squamous Cell Carcinoma of the Larynx Stage III; Squamous Cell Carcinoma of the Larynx Stage IV; Laryngeal Squamous Cell Carcinoma; Laryngectomy; Status; Laryngeal Cancer; Laryngeal Neoplasms
Keywords: induction chemotherapy; neoadjuvant treatment; immune checkpoint inhibitor; pembrolizumab; KEYNOTE; larynx organ preservation; laryngectomy-free survival; overall survival; event-free survival
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Laryngeal Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, open-label, controlled, two-armed parallel group, phase II multicenter larynx organ-preservation trial with randomization in a 1:1 ratio into standard arm vs. investigational arm with a flexible follow-up of 24-48 months
Masking Description: There will be no masking
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- A - Control (No Intervention): Standard-Arm:
  Short Induction (IC-1):
  T = Docetaxel 75 mg/m^2 i.v. day 1 P = Cisplatin 75 mg/m^2 i.v. day 1 Response evaluation will be performed in week 4 after IC-1 by endoscopic estimation of tumor-surface shrinkage (ETSS) to select nonresponders for early total laryngectomy (TL). Responders receive further 2 cycles TP followed by radiotherapy (RT) starting week 11.
  ETSS < 30% (Nonresponder):
  - TL + adjuvant RT or chemo-radiotherapy (CRT) according the decision of the tumor board
  ETSS >=30% (Responder):
  2 further TP cycles (IC-2 in week 5-7 and IC-3 in week 8-10; same doses as IC-1) Radiotherapy (RT) is accelerated IMRT with concomitant boost with total dose of 69.6 Gy applied over 5.5 weeks to all tumor localizations; clinically non-affected neck levels receive 51.6 Gy.
  * protocol is according exactly to the DeLOS-II protocol arm A in Dietz et al. Ann Oncol. 2018 Oct 1;29(10):2105-2114
- B - KEYTRUDA® (Experimental): Intervention arm aka Experimental-Arm:
  Treatment same as for patients randomized into the standard arm A + application of KEYTRUDA® (pembrolizumab), i.v., in 3-week cycle (q3w) 200 mg, starting day 1; for 17 cycles (12 months). Treatment with pembrolizumab will continue in the experimental arm regardless of ETSS status after IC-1 in both responders and laryngectomized nonresponders, independent from subsequent decision on adjuvant therapy after TL.
  Interventions: Biological: KEYTRUDA®

INTERVENTIONS:
Biological: KEYTRUDA® — 200 mg KEYTRUDA® i. v. in 3-week cycle (q3w)
  Other Names: Pembrolizumab; MK-3475
  Arms: B - KEYTRUDA®

SUMMARY:
ELOS is a prospective, randomized, open-label, controlled, two-armed parallel group, phase II multicentre trial in local advanced stage III, IVA/B head and neck squamous cell carcinoma of the larynx or hypopharynx (LHNSCC) with PD-L1-expression within tumor tissue biopsy, calculated as CPS ≥ 1 curable by total laryngectomy. Induction chemotherapy (IC) with Docetaxel and Cisplatin (TP) followed by radiation will be compared to additional PD-1 inhibition. Patients will be selected after short induction early response evaluation after the first cycle IC (IC-1) aiming on larynx organ-preservation by additional 2 cycles IC followed by radiotherapy (69.6 Gy) for responders achieving endoscopic estimated tumor surface shrinkage (ETSS) ≥ 30%. Nonresponders (ETSS < 30% or progressing disease) will receive total laryngectomy and selective neck dissection followed by postoperative radiation or chemoradiation according to the recommendation of the clinics multidisciplinary tumor board. However, Patients randomized into the intervention arm starting day 1 will receive 200 mg Pembrolizumab (MK-3475) i.v. in 3-week cycle (q3w) for 17 cycles (12 months). Treatment with pembrolizumab will continue in the experimental arm regardless of ETSS status after IC-1 in both responders and laryngectomized nonresponders, independent from subsequent decision on adjuvant therapy after TL.

DETAILED DESCRIPTION:
ELOS is a prospective, randomized, open-label, controlled, two-armed parallel group, phase II multicentre trial in local advanced stage III, IVA/B head and neck squamous cell carcinoma of the larynx or hypopharynx (LHNSCC) with PD-L1-expression within tumor tissue biopsy, calculated as CPS ≥ 1 curable by total laryngectomy. Induction chemotherapy (IC) with Docetaxel and Cisplatin (TP) followed by radiation will be compared to additional PD-1 inhibition. Patients will be selected after short induction early response evaluation after the first cycle IC (IC-1) aiming on larynx organ-preservation by additional 2 cycles IC followed by radiotherapy (69.6 Gy) for responders achieving endoscopic estimated tumor surface shrinkage (ETSS) ≥ 30%. Nonresponders (ETSS < 30% or progressing disease) will receive total laryngectomy and selective neck dissection followed by postoperative radiation or chemoradiation according to the recommendation of the clinics multidisciplinary tumor board. However, Patients randomized into the intervention arm starting day 1 will receive 200 mg Pembrolizumab (MK-3475) i.v. in 3-week cycle (q3w) for 17 cycles (12 months). Treatment with pembrolizumab will continue in the experimental arm regardless of ETSS status after IC-1 in both responders and laryngectomized nonresponders, independent from subsequent decision on adjuvant therapy after TL.

The primary objective of ELOS is to compare laryngectomy-free survival (LFS) achieved by adding KEYTRUDA® (pembrolizumab) to standard treatment and LFS after standard treatment according to the DeLOS-II protocol in advanced LHNSCC curable by laryngectomy.

Hypothesis: Adding PD-1 inhibition by pembrolizumab to organ-preservation chemoradiation treatment improves laryngectomy-free survival (LFS) compared to standard treatment according to the DeLOS-II protocol.

The secondary objectives are to compare Quality of Swallowing (QoS) assessed by FEES, event free survival (EFS) and overall survival (OS) achieved by adding KEYTRUDA® (pembrolizumab) to standard treatment and QoS, EFS and OS after standard treatment according to the DeLOS-II protocol in advanced LHNSCC. In general, the main interest in trials focusing on improving quality and degree of larynx organ preservation is late functional (in particular "swallowing") outcome. Current instruments assessing hrQoL are less meaningful than direct objective assessment of swallowing utilizing physical examination like FEES. FEES is a well approved and reliable method and allows clear scoring of quality of swallowing for instance by applying the Rosenbek Scale. Therefore, the investigators decided to avoid any questionnaires for this assessment including those approved for use in head and neck cancer, as they fail to specifically address the main study outcome, functional larynx organ preservation.

Hypothesis: Adding PD-1 inhibition by KEYTRUDA® (pembrolizumab) to organ-preservation chemoradiation treatment improves QoS, EFS and OS compared to standard treatment according to the DeLOS-II protocol. EFS events are defined as any event either in interfering with proper larynx organ function (independent of the cause, tumor- or treatment related), relapse (local, loco-regional, or distant), or death.

ELIGIBILITY:
Inclusion Criteria:

Participants are eligible to be included in the study only if all of the following criteria apply:

1. Male and female participants who are at least 18 years of age on the day of signing informed consent with histologically confirmed diagnosis of squamous cell carcinoma (SCC) of the larynx or hypopharynx according to the decision of the multidisciplinary tumor board suitable for total laryngectomy can be enrolled in this study.
2. Stage III, IVA or IVB, whenever clear resection margins R0 >5 mm can be achieved and no radiologic signs of extranodal extension of neck nodes are present.
3. Have provided newly obtained excisional biopsy of a tumor lesion not previously irradiated. Formalin-fixed, paraffin embedded (FFPE) tissue blocks are preferred to slides.
4. PD-L1-expression* within the tumor biopsy, CPS ≥1
5. Male participants:

   A male participant must agree to use a contraception as detailed in Appendix 3 of this protocol during the treatment period and for at least 120 days after the last dose of study treatment and refrain from donating sperm during this period.
6. Female participants:

   A female participant is eligible to participate if she is not pregnant (see Appendix 3), not breastfeeding, and at least one of the following conditions applies:
   1. Not a woman of childbearing potential (WOCBP) OR
   2. A WOCBP who agrees to follow the contraceptive guidance during the treatment period and for at least 120 days after the last dose of study treatment.
7. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1. Evaluation of ECOG is to be performed within 7 days prior to the date of allocation/randomization.
8. Have adequate organ function as defined in the (Table 4) of the protocol. Specimens must be collected within 10 days prior to the start of study treatment.

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

1. A WOCBP who has a positive urine pregnancy test within 72 hours prior to receiving the first dose of study medication (see Appendix 3). If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
2. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti PD L2 agent or with an agent directed to another stimulatory or co-inhibitory receptor on T or NK cells (e.g., CTLA-4, OX 40, CD137).
3. Has received prior systemic anti-cancer therapy including investigational agents.
4. Has received prior radiotherapy.
5. Has received a live vaccine or live-attenuated vaccine within 30 days prior to the first dose of study drug. Administration of killed vaccines is allowed.
6. Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study intervention.
7. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
8. Has a history of a second malignancy, unless potentially curative treatment has been completed with no evidence of malignancy for 2 years.
9. Has known distant metastases including active CNS metastases and/or carcinomatous meningitis.
10. Has severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients.
11. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment and is allowed.
12. Has a history of (non-infectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease.
13. Has an active infection requiring systemic therapy.
14. Has a known history of Human Immunodeficiency Virus (HIV) infection. Note: No HIV testing is required unless mandated by local health authority.
15. Has a known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as HCV RNA [qualitative] is detected) infection. Note: no testing for Hepatitis B and Hepatitis C is required unless mandated by local health authority.
16. Has a known history of active TB (Bacillus Tuberculosis).
17. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
18. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
19. Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment.
20. Has had an allogenic tissue/solid organ transplant.
21. Has a known intolerance to one of the substances administered during treatment including e.g. antibiotics, antiemetics, etc. or any other component of concurrent auxiliary medication.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2024-04-17 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
laryngectomy-free survival (LFS) | 24 to 48 months (flexible follow-up)
  Laryngectomy-free survival (LFS) is the survival of the patient with larynx at place aka survival without laryngectomy, in the intent-to-treat population (follow-up of the total cohort until 24 months after randomization of the last patient accrued). Laryngectomy or death from any cause count as event.
  We measure LFS in the intent-to-treat population as the survival time of patients with larynx at place, which is the time interval from date of randomization until date of LFS event (follow-up of the total cohort until 24 months after randomization of the last patient accrued). Laryngectomy or death from any cause count as LFS event. Patients lost to follow-up will be censored at date of last visit with larynx at place. Recruitment will be over 2 years and all patients will be followed up for at least 2 years, resulting in a maximum follow-up time of 4 years.

SECONDARY OUTCOMES:
overall-survival (OS) | 24 to 48 months (flexible follow-up)
  Overall survival (OS) is the survival of the patient without death from any cause, in the intent-to-treat population (follow-up of the total cohort until 24 months after randomization of the last patient accrued).
  We measure OS in the intent-to-treat population as the survival time of patients as the time interval from date of randomization until date of death from any cause (follow-up of the total cohort until 24 months after randomization of the last patient accrued). Patients lost to follow-up will be censored at date of last visit. Recruitment will be over 2 years and all patients will be followed up for at least 2 years, resulting in a maximum follow-up time of 4 years.
quality of swallowing (QoS) and freedom from laryngoesophageal dysfunction (FFLED) | 24 to 48 months (flexible follow-up)
  QoS will be assessed by fiber-endoscopic estimation of swallowing (FEES) at time of randomization and 6 and 24 months after first cycle induction chemo using the Rosenbek Scale (RS). De novo dysphagia (RS for aspiration and airway invasion/penetration >1) or exacerbation of existing dysphagia RS 2-5 to RS ≥6 (aspiration), is loss of freedom from laryngo-esophageal dysfunction (FFLED; event). An event might also be persistence of either tracheostoma or gastric tube at 24 months (event at 24 months) or total laryngectomy or death from any cause.
  We measure FFLED in the intent-to-treat population as time interval from date of randomization until date of event (follow-up of the total cohort until 24 months after randomization of the last patient accrued). Patients lost to follow-up will be censored at date of last visit without event. Recruitment will be over 2 years and all patients will be followed up for at least 2 years, resulting in maximum follow-up of 4 years.
event-free survival (EFS) | 24 to 48 months (flexible follow-up)
  Event-free survival (EFS) is the survival of the patient without any event. Total laryngectomy (TL), progressing disease, occurrence of new lesions, local or nodal relapse, distant metastases or death from any cause count as event.
  We measure EFS in the intent-to-treat population as the time interval from date of randomization until date of any event (follow-up of the total cohort until 24 months after randomization of the last patient accrued). Patients lost to follow-up will be censored at date of last visit without event. Recruitment will be over 2 years and all patients will be followed up for at least 2 years, resulting in a maximum follow-up time of 4 years.
event-free survival (EFS), alternative definition | 24 to 48 months (flexible follow-up)
  Event-free survival (EFS) is the survival of the patient without any event. As early total laryngectomy (TL) of nonresponders with ETSS <30% assessed by early response evaluation in week 4 is per-protocol therapy of LHSCC patients, which according to insufficient response to IC-1 cannot be selected for further 2 cycles TP followed by RT to achieve larynx organ-preservation, the alternative analysis of EFS will not consider early TL of nonresponders as event. However, progressing disease, occurrence of new lesions, local or nodal relapse, distant metastases or death from any cause and TL >2 months after IC-1 or loss of FFLED count as event.
  We measure EFS in the intent-to-treat population as the time interval from date of randomization until date of event. Patients lost to follow-up will be censored at date of last visit without event. Recruitment will be over 2 years and all patients will be followed up for at least 2 years, resulting in a maximum follow-up time of 4 years.

CONTACTS AND LOCATIONS:
Locations (9):
- Germany (9):
  - Universitätsklinikum Mannheim, Klinik für Hals-Nasen-Ohrenheilkunde Theodor-Kutzer-Ufer 1-3, Mannheim, Baden-Würtemberg
  - Universitätsklinikum Ulm / Ulm University Medical Center, Klinik für Hals- Nasen-Ohrenheilkunde und Kopf-Halschirurgie, Frauensteige 12, Ulm, Baden-Würtemberg
  - Klinikum rechts der Isar der TU München, Klinik und Poliklinik für Hals-, Nasen- und Ohrenheilkunde, Ismaninger Straße 22, München, Bavaria
  - Universität Regensburg, Klinik und Poliklinik für Strahlentherapie Franz-Josef-Strauss-Allee 11, Regensburg, Bavaria
  - Universitätsklinikum Würzburg, Klinik für Hals-, Nasen-, Ohrenheilkunde, Josef-Schneider-Straße 8, Würzburg, Bavaria
  - Klinikum Ernst von Bergmann, Klinik für Hämatologie, Onkologie und Palliativmedizin, Charlottenstr. 72, Potsdam, Brandenburg
  - Universitätsklinikum Köln, Klinik für Hals-, Nasen-, Ohrenheilkunde, Kerpener Str. 62, Cologne, North Rhine-Westphalia
  - University of Leipzig, Department für Kopf- und Zahnmedizin, Klinik und Poliklinik für Hals-, Nasen- und Ohrenheilkunde, Liebigstrasse 12, Leipzig, Saxon
  - Universitätsklinikum Jena Klinik für Hals-, Nasen- und Ohrenheilkunde, Am Klinikum 1, Jena, Thuringia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dietz A, Wichmann G, Kuhnt T, Pfreundner L, Hagen R, Scheich M, Kolbl O, Hautmann MG, Strutz J, Schreiber F, Bockmuhl U, Schilling V, Feyer P, de Wit M, Maschmeyer G, Jungehulsing M, Schroeder U, Wollenberg B, Sittel C, Munter M, Lenarz T, Klussmann JP, Guntinas-Lichius O, Rudack C, Eich HT, Foerg T, Preyer S, Westhofen M, Welkoborsky HJ, Esser D, Thurnher D, Remmert S, Sudhoff H, Gorner M, Bunzel J, Budach V, Held S, Knodler M, Lordick F, Wiegand S, Vogel K, Boehm A, Flentje M, Keilholz U. Induction chemotherapy (IC) followed by radiotherapy (RT) versus cetuximab plus IC and RT in advanced laryngeal/hypopharyngeal cancer resectable only by total laryngectomy-final results of the larynx organ preservation trial DeLOS-II. Ann Oncol. 2018 Oct 1;29(10):2105-2114. doi: 10.1093/annonc/mdy332. PMID 30412221
- [Background] Bindewald J, Herrmann E, Dietz A, Wulke C, Meister E, Wollbruck D, Singer S. [Quality of life and voice intelligibility in laryngeal cancer patients--relevance of the "satisfaction paradox"]. Laryngorhinootologie. 2007 Jun;86(6):426-30. doi: 10.1055/s-2007-966167. German. PMID 17654777
- [Background] Rosenbek JC, Robbins JA, Roecker EB, Coyle JL, Wood JL. A penetration-aspiration scale. Dysphagia. 1996 Spring;11(2):93-8. doi: 10.1007/BF00417897. PMID 8721066
- [Derived] Wichmann G, Wald T, Pirlich M, Napp J, Munter I, Asendorf T, Tostmann R, Vogt J, Vogel K, Meuret S, Stoehr M, Zebralla V, Nicolay NH, Kuhnt T, Hambsch P, Guntinas-Lichius O, Klussmann JP, Wiegand S, Dietz A. The European Larynx Organ Preservation Study [MK-3475-C44]. Front Oncol. 2024 Aug 22;14:1433238. doi: 10.3389/fonc.2024.1433238. eCollection 2024. PMID 39239277